CLINICAL TRIAL: NCT02070562
Title: Human Milk Profiles and Dietary Intake of Chinese Lactating Mothers During Early Lactation Period in Shanghai
Acronym: MuRu
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dumex Baby Food Co., Ltd. (Industry)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HMR.1.C/A
Record Dates: First submitted 2014-01-27; First posted 2014-02-25 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Breast Milk
Keywords: breast milk, dietary survey

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breast milk from 0-42 days postpartum

GROUPS / COHORTS (2):
- Community Group: Chinese lactating mothers from community maternal & child healthcare centre
- VIP Group: Chinese lactating mothers from VIP clinics (maternal care center)

SUMMARY:
This study aims to investigate breast milk composition and dietary habits of Chinese lactating mothers. Further understanding of the composition of human milk will help to understand the nutritional needs of mothers and their infants in their early phase of life which eventually will help to support breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy mothers who give birth to a healthy term infant (37-42 weeks) whose birth weight is >10 and <90 percentiles gestational birth weight chart.
* Aged 20 - 40 years.
* Mothers who intend to exclusively breastfeed the infant for more than 6 weeks.
* Chinese ethnicity, including both parents.
* Mothers who sign the informed consent form in writing.

Exclusion Criteria:

Mothers:

* Participation in any other studies involving investigational or marketed products concomitantly or two weeks prior to entry into the study.
* Difficult to follow up and/or locate (e.g. known transfer to other hospitals, residing outside Shanghai, plan to move out of Shanghai).
* Current smoker or having smoked during the pregnancy.
* Having consumed alcoholic drinks during pregnancy or lactation.
* Illegal drug abuser: cannabinoids (marijuana, hashish), stimulants (cocaine, amphetamine, methamphetamine), opioid (heroin, opium).
* Acute infection disease or neoplastic disease or any kind of weakening or debilitating conditions (no history of positive HBV, HCV or HIV serological test at any time during the pregnancy).
* Use of drug or pharmacologically active substances (e.g. herbal products, traditional medicine) to treat a particular disease or medical condition from the beginning of lactation ( those who consume herbal/traditional medicine for maintaining or improving well-being will still be included).
* Presence of mastitis, fungal infections of the nipple or areola; reactivation of herpes simplex (HSV) or varicella zoster infection in the mammary or thoracic region at the time of enrolment.
* Presence of endocrinology diseases, particularly diabetes mellitus and gestational diabetes.
* Presence of obesity (pre-pregnancy BMI > 28).
* Presence of chronic diseases such as cardiovascular, renal, respiratory and hepatic diseases.
* Presence of psychosis and severe post-partum depression.
* Presence of autoimmune disease such as systemic lupus erythematosus, systemic scleroderma, ulcerative colitis, Crohn's disease, celiac disease.
* Women whose health condition, according to the investigator's judgement, could interfere with the study conduct and assessment.
* Mothers who have given birth to twins or multiples or infant conceived with Assisted Reproductive Technology (ART).
* Elimination diet due to chronic allergic diseases or vegan.
* Incapability of subject to comply with study protocol or investigator's uncertainty about the willingness or ability of the mothers to understand and comply with the protocol requirements.

Infants:

* Any congenital abnormality, chromosomal disorder or severe disease which could interfere with the study conduct and assessment.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General health lactating mothers
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-08 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Breast milk composition | 0-42 day postpartum
  Human milk oligosaccharides profiles, fatty acids profile, macronutrients and energy content will be measured.

SECONDARY OUTCOMES:
Growth | 0-42 day postpartum
  Infant's anthropometrics (weight, length, head circumference).
Maternal diet survey | 0-42 day postpartum
  Dietary macronutrients and energy intake, and food patterns will be assessed.
Infection | 0-42 day postpartum
  Parent-reported infection patterns of infants during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, professor, Principal Investigator — Shanghai Children's Medical Center Affiliated Shanghai Jiao Tong University, School of Medicine
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China